CLINICAL TRIAL: NCT01345110
Title: A Longitudinal Population Study on Brain Aging and Mental Performances for the 1935-1939 Born People Living in Abbiategrasso (a Small Town Near Milan)
Brief Title: A Longitudinal Multidimensional Population Study on Brain Aging
Acronym: InveCeAb
Status: Completed | Type: Observational
Sponsor: Fondazione Golgi Cenci (Other)
Collaborators: Alzheimer Federation Italy (Other); Mario Negri Institute for Pharmacological Research (Other); University of Pavia (Other); Camillo Golgi Geriatric Institute (Other)
Responsible Party: Principal Investigator, Antonio Guaita, MD, director, Fondazione Golgi Cenci
Other Study IDs: 01
Record Dates: First submitted 2011-04-21; First posted 2011-04-29 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Dementia; Alzheimer Disease; Vascular Dementia
Keywords: dementia; mild cognitive impairment; prevalence; incidence; elderly; longitudinal study; population study
MeSH Terms: conditions — Dementia; Alzheimer Disease; Dementia, Vascular; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood and serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Longitudinal observational study of cognitive functions, physical health and biological parameters in the whole population living in Abbiategrasso born between 1935 and 1939,1773 subjects, followed for six years in order to know the prevalence and the incidence of dementia and risk and protective factors of normal and pathological mental aging.

The peculiarities of this study that must assure the outcome efficacy are:

* Selected age: since 70-75 years old people represents a transition age from adulthood to old age, it is of special interest to study the evolution of psychic and physical functions of this population
* Whole population not a sample study
* Location: the small area involved (Abbiategrasso is a town of 30.000 inhabitants)can contribute to guarantee more homogeneity among the subjects and reduce undesired variability
* multidimensional assessment(biological, clinical, social, psychological data collected) After initial screening, the recruited population will be followed up for two more times (every two years )

DETAILED DESCRIPTION:
Background:

Dementia is one of the most troubling neurodegenerative syndrome whose prevalence and incidence is strongly increasing. The etiology and physiopathology of the process that causes dementia are still controversial and largely unknown. So it is of paramount importance to isolate risk and protection factors related to dementia syndrome and Alzheimer disease. These meager known factors (biological, as well as social and neuropsychological) can be better investigated through a multidimensional longitudinal study in a homogeneous population by age and place.

Method:

People belonging to the selected population (1773 subjects living in Abbiategrasso and born between 1935 - 1939) were invited to participate at a comprehensive assessment which was divided in two appointments:

* a first appointment (about 1 hour and half) for blood sample, social questionnaire, anthropometric and walking speed evaluation ;
* a second one (2 hours)for clinical examination and neuropsychological assessment of mood and cognitive function.

Recruitment. People were recruited through several steps:

* involvement of the family doctor;
* a general call, based on age group(1935,1936, 1937, 1938, 1939), since to be born in the same year is an identity mark for these generations;
* kick-off meetings for each age class explaining aims and methods of the research, followed by a party with music, plays and some lotteries
* a letter with the date of the appointment followed by the phone call whenever the phone number is available
* further letters and call until either a rejection or an appointment was taken.

Assessment. Professionals and instruments:

* Trained interviewers, one social worker and two nurses, administer the social questionnaire that is partly derived from the CERAD and from other longitudinal studies.
* Trained psychologists administer a neuropsychological battery exploring mood (GDS 15 items), verbal and visual memory (Rey 15-item Memory Test, and the Rey-Osterrieth Complex Figure Test (ROCF) recall; Babcock Story Recall Test ), executive function ( TMTA and TMTB; copy of ROCF), attention (Numerical Attention), abstract reasoning (Raven's Coloured Progressive Matrices), screening cognitive test (Clock test and MMSE).
* Clinical interview and visit are executed by expert geriatricians, members of the same geriatric staff who apply diagnostic criteria for dementia (DSM IV), Alzheimer disease (NINCDS ADRDA diagnostic criteria); Vascular dementia (NINDS -AIREN criteria); Lewy Body dementia (third report, DLB consortium); frontotemporal dementia ( 2002 modified Consensus conference criteria). Other cognitive problems were classified as Mild Cognitive Impairment (MCI) following Petersen's criteria or Cognitive Impairment No Dementia (CIND) when cognitive impairments are in areas other than memory and they do not meet whole criteria for dementia. Every diagnostic conclusion is revised by another doctor; in case of discrepancies a third geriatrician, chief of the study, intervenes to arbitrate.

All the instruments were pre tested for inter rater reliability in a similar population attending a geriatric day hospital, and some general agreement sessions were performed before and during the screening.

ELIGIBILITY:
Inclusion Criteria:

* to be resident in Abbiategrasso
* to be born between 1935 and 1939

Exclusion Criteria:

* to refuse to participate
* te be not contactable in any way (mail, telephone)
* to be legally resident, but actually living somewhere else

Ages: 70 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All the 1773 residents of Abbiategrasso, a town of 30.000 inhabitants near Milan, Lombardy, Italy, born from 1935 to 1939 : 1724 subjects meets the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 1321 (Actual)
Dates: Start 2009-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The proportion of the recruited persons who will develop Dementia syndrome, Alzheimer disease, Vascular dementia, Lewy Body dementia, frontotemporal dementia, Mild Cognitive Impairment, Cognitive Impairment No Dementia | six years
  These are the criteria used for the definitions :
  * DSM IV for Dementia syndrome
  * NINCDS ADRDA diagnostic criteria for Alzheimer disease
  * NINDS -AIREN criteria for Vascular dementia
  * Third report, DLB consortium for Lewy Body dementia
  * 2002 modified Consensus Conference criteria for frontotemporal dementia
  * Report of the MCI Working Group of the European Consortium on Alzheimer's Disease for Mild Cognitive Impairment (MCI)
  * Absence of the first criteria for MCI (subjective complain) for the definition of Cognitive Impairment No Dementia (CIND)

SECONDARY OUTCOMES:
The proportion of persons who will exhibit a performance decrease equal or more than of 1,5 standard deviation of the mean in the reference population in screening cognitive tests or in memory tests (verbal and visual memory) or in executive tests | six years
  * Screening cognitive tests: Clock test and MMSE.
  * Memory tests: Babcock Story Recall Test , Rey 15-item Memory Test, and the Rey-Osterrieth Complex Figure Test (ROCF) recall.
  * Executive tests:Trial making A and B; copy of ROCF
Neuropsychological baseline features of the persons who will develop dementia or cognitive impairment | six years
  * Mood: GDS 15 items
  * Verbal and visual memory: Babcock Story Recall Test, Rey 15-item Memory Test, and the Rey-Osterrieth Complex Figure Test (ROCF) recall
  * Executive function: TMTA and TMTB; copy of ROCF
  * Attention: Numerical Attention
  * Abstract reasoning: Raven's Coloured Progressive Matrices
  * Screening cognitive test: Clock test and MMSE
Clinical baseline features of the persons who will develop dementia or cognitive impairment | six years
  * Index of co morbidities as defined by CIRS (Cumulative Index Rating Scale)
  * Standard neurological examination
Social baseline features of the persons who will developed dementia or cognitive impairment | six years
  * Stressful life events as defined in GALES (Geriatric Adverse Life Event Scale)
  * Physical activity
  * Social network
Genetic baseline features of the persons who will developed dementia and/or cognitive impairment | six years
  * ApoE
  * Inflammatory cytokines

CONTACTS AND LOCATIONS:
Overall Officials: ANTONIO GUAITA, MD, Study Director — Golgi Cenci Foundation (research and study on aging)
Locations (1):
- Golgi Cenci Foundation, Abbiategrasso, Milan, Italy

REFERENCES:
- [Background] Guaita A, Forloni GL, Ferretti V, Villani S, Fossi S, Colombo M, Salvini Porro G InveCe.Ab: a multidimensional population study on brain aging for the 1935 - 1939 born people in a small town near Milan JNHA ( the Journal of Nutrition, Health &Aging) 2010; 14 (supplement 2): S17
- [Background] Guaita A, Colombo M, Vaccaro R, Fossi S, Vitali SF, Forloni G, Polito L, Davin A, Ferretti VV, Villani S. Brain aging and dementia during the transition from late adulthood to old age: design and methodology of the "Invece.Ab" population-based study. BMC Geriatr. 2013 Sep 24;13:98. doi: 10.1186/1471-2318-13-98. PMID 24063518
- [Background] Guaita A, Vaccaro R, Davin A, Colombo M, Vitali SF, Polito L, Abbondanza S, Valle E, Forloni G, Ferretti VV, Villani S. Influence of socio-demographic features and apolipoprotein E epsilon 4 expression on the prevalence of dementia and cognitive impairment in a population of 70-74-year olds: the InveCe.Ab study. Arch Gerontol Geriatr. 2015 Mar-Apr;60(2):334-43. doi: 10.1016/j.archger.2014.11.006. Epub 2014 Nov 25. PMID 25466513
- [Derived] Valla LG, Rossi M, Gaia A, Guaita A, Rolandi E. The Impact of the COVID-19 Pandemic on Oldest-Old Social Capital and Health and the Role of Digital Inequalities: Longitudinal Cohort Study. J Med Internet Res. 2025 Jan 9;27:e62824. doi: 10.2196/62824. PMID 39784108
- [Derived] Rolandi E, Rossi M, Colombo M, Pettinato L, Del Signore F, Aglieri V, Bottini G, Guaita A. Lifestyle, Cognitive, and Psychological Factors Associated With a Resilience Phenotype in Aging: A Multidimensional Approach on a Population-Based Sample of Oldest-Old (80+). J Gerontol B Psychol Sci Soc Sci. 2024 Oct 1;79(10):gbae132. doi: 10.1093/geronb/gbae132. PMID 39096236
- [Derived] Rolandi E, Zaccaria D, Vaccaro R, Abbondanza S, Pettinato L, Davin A, Guaita A. Estimating the potential for dementia prevention through modifiable risk factors elimination in the real-world setting: a population-based study. Alzheimers Res Ther. 2020 Aug 7;12(1):94. doi: 10.1186/s13195-020-00661-y. PMID 32767997
- See also: official web site of the organization responsible for the study — http://www.golgicenci.it
- See also: official website of the caregivers organization, partner in the sponsorship of the research — http://www.alzheimer.it